CLINICAL TRIAL: NCT00409786
Title: Virtual Lifestyle Management: Prevention Through the UPMC Patient Portal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Air Force Office of the Surgeon General (U.S. Federal Agency)
Responsible Party: Kathleen McTigue, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 0606089; W81XWH-04-2-0030
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Results first posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Obesity
Keywords: Obesity; Diabetes; Internet; Obesity with high cardiovascular risk
MeSH Terms: conditions — Obesity; Diabetes Mellitus

INTERVENTIONS:
Behavioral: Virtual Lifestyle Management (VLM) — 16 weekly lessons followed by monthly maintenance lessons

SUMMARY:
Diabetes affects 18 million Americans and costs over $132 billion in both direct treatment and lost productivity per year. It is known that weight loss, improved diet and increased exercise can result in improvement in glucose, lipid, and blood pressure control in patients with diabetes and reduce the incidence of diabetes in individuals at high risk. Effective delivery of proven, comprehensive lifestyle programs is difficult because of associated high costs.

The internet provides a venue to deliver these lifestyle programs to large numbers of individuals while decreasing the cost per person. HealthTrak, the University of Pittsburgh Medical Center (UPMC) patient portal, provides an ideal setting to test such a program. HealthTrak provides participants with access to individual medical information while facilitating electronic communication with their physicians. Portal enhancements will allow the delivery of a comprehensive lifestyle intervention aimed at weight loss, improved diet, and increased exercise, and provide the opportunity to communicate with experts regarding concerns.

Through this project, we will evaluate the modification of a successful comprehensive lifestyle intervention for delivery through HealthTrak. We will enroll and follow 50 individuals with diabetes or at high risk for diabetes for 12 months and examine change in parameters including diet, weight, physical activity, hemoglobin A1C, glucose, blood pressure, and lipid profile.

DETAILED DESCRIPTION:
Diabetes affects 18 million Americans and costs over $132 billion in both direct treatment and lost productivity per year. It is known that weight loss, improved diet and increased exercise can result in improvement in glucose, lipid, and blood pressure control in patients with diabetes and reduce the incidence of diabetes in individuals at high risk. Effective delivery of proven, comprehensive lifestyle programs is difficult because of associated high costs.

The internet provides a venue to deliver these lifestyle programs to large numbers of individuals while decreasing the cost per person. HealthTrak, the University of Pittsburgh Medical Center (UPMC) patient portal, provides an ideal setting to test such a program. HealthTrak provides participants with access to individual medical information while facilitating electronic communication with their physicians. Portal enhancements will allow the delivery of a comprehensive lifestyle intervention aimed at weight loss, improved diet, and increased exercise, and provide the opportunity to communicate with experts regarding concerns.

Through this project, we will evaluate the modification of a successful comprehensive lifestyle intervention for delivery through HealthTrak. We will enroll and follow 50 individuals with diabetes or at high risk for diabetes for 12 months and examine change in parameters including diet, weight, physical activity, hemoglobin A1C, glucose, blood pressure, and lipid profile

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI≥25) and one of the following:

Hypertension, Diabetes, glucose intolerance, dyslipidemia

* Age 18-80
* Agrees to participate in the Virtual Lifestyle Management (VLM) program and evaluation
* Computer access to UPMC Health Trak
* Regular access to a scale

Exclusion Criteria:

* Pregnancy
* Inability to participate in moderate exercise as determined by the primary care physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hess, MD, MSc, Principal Investigator — University of Pittsburgh Medical Center; Kathleen McTigue, MD, MSc, Study Director — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527

RESULTS

PARTICIPANT FLOW:
Groups:
- VLM Online Lifestyle Counseling: Overweight primary care patient participants receiving the Virtual Lifestyle Management (VLM) Program online lifestyle counseling intervention.
Period: Overall Study
Arm/Group | VLM Online Lifestyle Counseling
Started | 50
Completed | 47
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | VLM Online Lifestyle Counseling
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 51.94 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Time Frame: Baseline and 1 year
Population: Of the original 50 participants, 12 month data was collected for 45 (90%) of them. Analysis was conducted on those participants with 12 month data.
Measure: Mean (95% Confidence Interval); unit: kg
Groups:
- Group 1: All participants
Arm/Group | Group 1
Number analyzed (Participants) | 45
kg | -4.79 [-7.36 to -2.22]

2. Secondary Outcome: Blood Pressure
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Lipid
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: A1C (if Applicable)
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Fat Consumption
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Health Related Quality of Life
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Physical Activity
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | VLM Online Lifestyle Counseling
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No